CLINICAL TRIAL: NCT01364506
Title: Randomized Clinical Study of the Effects of Aerobic Water Exercise on Maternal Cardiovascular Adaptation to Pregnancy
Brief Title: The Effects of Aerobic Water Exercise on Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UPECLIN HC FM Botucatu Unesp (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government); Federal University of São Paulo (Other); Faculdade de Medicina de Botucatu, UNESP, Botucatu, Brasil (Other)
Responsible Party: Iracema de Mattos Paranhos Calderon, Department of Gynecology and Obstetrics of Botucatu Medical School - São Paulo State University/UNESP. Botucatu, Brazil
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: upeclin/HC/FMB-Unesp-54
Record Dates: First submitted 2011-05-31; First posted 2011-06-02 (Estimated); Last update posted 2011-06-02 (Estimated); Status verified 2011-05

CONDITIONS: Pregnancy Related; Physical Activity
Keywords: Cardiovascular capacity; Water exercise; Hydrokinetic Therapy; Pregnancy; Perinatal outcomes
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Water exercise (Experimental)
  Interventions: Other: Water aerobic exercise
- Control (No Intervention)

INTERVENTIONS:
Other: Water aerobic exercise — The hydrotherapy program of Prevedel et al.14 was used. One-hour sessions, led by a physiotherapist under the supervision of an obstetrician, were held three times a week in an indoor swimming-pool heated at 28oC-32oC, and consisted of exercises of moderate intensity (60-70% of maximum heart rate). Subgroups of up to 10 subjects participated in each session. Sessions were offered at different times of the day (morning, afternoon, and evening).
  The exercises included 5 phases: stretching, warm up, endurance training, strength training and relaxation with breathing exercises, in accordance with the recommendations of ACOG11.
  Arms: Water exercise

SUMMARY:
Objective: To assess the relationship between maternal cardiovascular capacity and aerobic water exercise during the gestational periods of hemodynamic overload. Study design: randomized clinical trial, with 41 healthy pregnant women assigned to one of two groups: Control and Water exercise. Maternal cardiovascular capacity (maximum oxygen consumption, cardiac output, stroke volume, heart rate and mean arterial pressure), physical performance (relative HR, treadmill speed and self-perceived exertion) and neonatal outcome (gestational age, weight, Apgar index and length of infant's hospitalization) were assessed. Means were evaluated by dependent and independent t-tests, and proportions by the chi-square method (p<0.05). Results: The control variables showed that the groups were homogeneous. Water exercise was associated with maintenance of VO2max, increase in stroke volume and cardiac output, and better performance on stress tests in the third trimester of gestation. No significant difference in neonatal variables was observed. Conclusion: Water exercise maintained cardiovascular capacity and performance under submaximal stress, and did not affect hemodynamic adaptation to gestation or neonatal outcome.

DETAILED DESCRIPTION:
INTRODUCTION

Significant hemodynamic changes take place during the short period of pregnancy, very often placing a major burden on the maternal cardiovascular system. Normal pregnancy is characterized by an increase in cardiac output (CO), stroke volume (SV), heart rate (HR) and blood volume, and decrease in arterial pressure and vascular resistance. Classic studies have demonstrated an increase of up to 50% in maternal CO during the second and third trimesters. These circulatory adaptations are responsible for supplying nutrients and oxygen to the placenta and the fetus.

The physiological changes that follow regular exercise improve training efficiency and performance, defining the concept of adaptation to exercise or aerobic training. Exercise causes the heart and lungs to be more efficient by increasing cardiovascular capacity or resistance. CO, SV and maximum oxygen consumption (VO2max) increase while HR and AP decrease. The importance of these effects on overall health has been recognized by the most outstanding medical and scientific groups. Therefore, regular exercise has been widely promoted and a large number of women decide to begin or continue to exercise during pregnancy.

This change in women's behavior has become a matter of concern among obstetricians and has important practical implications - is the maternal body apt to bear the hemodynamic burden of pregnancy in association with exercise stress? Studies on the effects of exercise on pregnancy are scarce and show conflicting results, probably due to differences in exercise frequency, intensity, type, duration, and gestational age at training initiation.

Aiming at standardizing exercise practice and thus promote materno-fetal health, the American College of Obstetricians and Gynecologists (ACOG) issued, in 1985, guidelines for exercise during pregnancy. In subsequent reviews, new recommendations were added, and water exercise during pregnancy was recommended.

Water exercise offers some particular benefits that include the maintenance of body temperature, control of gestational edema, and increase in diuresis. Moreover, it can be easily performed up to the end of pregnancy, which favors compliance. These advantages added to the fact that it has no adverse effect on the fetus explain the preference for this kind of exercise during pregnancy.

Considering the lack of scientific evidence of the effects of exercise during pregnancy, and the results obtained in our previous work, the purpose of this study was to assess the relationship of aerobic water exercise during the gestational periods of greater hemodynamic burden with maternal cardiovascular capacity and neonatal outcomes.

METHODS

This study is part of a project approved by the Committee of Research Ethics of the Botucatu Medical School-UNESP on May 10, 1999.

Study design: randomized clinical, without intention to treat. Study subjects: All the eligible women who volunteered to participate were sequentially enrolled and randomized to one of two groups according to a computer-generated randomization list of numbers created with Epi-Info software. Each sequential number corresponded to a sealed opaque envelope containing the information on the randomization group in order to ensure concealment. Group 1 consisted of 29 women engaged in Water Exercise, and group 2 included 31 pregnant women not participating in the program (control). Variables: the independent variable studied was the practice of water exercise. The control variables, which were assessed at baseline, included age, parity, pre-gestational body mass index (BMI), HR and MAP, smoking, sedentarism, and gestational age at baseline and at stress testing. The dependent variables regarding cardiovascular capacity and physical performance at the submaximal stress test were VO2max; SV; CO; HR and MAP, relative HR treadmill speed and scores obtained with the scale of Borg. Neonatal variables included gestational age, weight; Apgar index at minute 1 and at minute 5, and length (days) of infant's hospitalization.

Assessment of cardiovascular capacity: performed during prenatal visits at 16-20, 28-33 and 34-39 weeks. Cardiovascular capacity was evaluated by using a treadmill submaximal stress test, according to the protocol of Balke-Ware & Bruce that requires five minutes on treadmill at fixed incline and constant individualized speed with AP and HR monitoring. Assessment of physical performance at stress testing - for this purpose, relative HR, treadmill speed and the Borg scale scores, obtained during testing, were used. A specific questionnaire was administered to all subjects in order to quantify stress perception during testing.

Data processing and analyses - given that the aim of this study was to assess the efficacy (exploratory and not intention-to-treat) of water exercise during pregnancy, our analysis included only the subjects who underwent cardiovascular assessment at the three study moments and missed no more than 2 exercise sessions/month. These data were stored in a specific database Statistical analysis was performed with SPSS software version 10.0.7. Means were compared using ANOVA followed by t-tests for independent (between groups) and dependent (within groups) samples. Data were adequately transformed when necessary. Proportions were compared by the chi-square test (X2). Statistical significance was set at 5% (p<0.005).

ELIGIBILITY:
Inclusion Criteria:

* Low-risk (healthy) pregnant women
* At 16-20 weeks of gestation
* Seen at the Prenatal Care Service for Low-risk Pregnancies of Botucatu Medical School-UNESP

Exclusion Criteria:

* Twin pregnancy
* Clinical or obstetric disorder contraindicating an exercise program
* Withdrawal from prenatal care at our service
* Loss to follow-up; and failure to attend three (or more) exercise sessions, which was considered non-compliance to the aerobic water exercise program

Ages: 15 Years to 26 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 41 (Actual)
Dates: Start 2000-01; Primary Completion 2001-04 (Actual); Study Completion 2001-04 (Actual)

PRIMARY OUTCOMES:
Cardiovascular capacity | 39 weeks
  Performed during prenatal visits at 16-20, 28-33 and 34-39 weeks. Cardiovascular capacity was evaluated by using a treadmill submaximal stress test, according to the protocol of Balke-Ware & Bruce that requires five minutes on treadmill at fixed incline and constant individualized speed with AP and HR monitoring.

SECONDARY OUTCOMES:
Assessment of physical performance at stress testing; stress perception during testing | 39 weeks
  Relative HR, treadmill speed and the Borg scale scores, obtained during testing, were used. A specific questionnaire was administered to all subjects in order to quantify stress perception during testing.

CONTACTS AND LOCATIONS:
Overall Officials: Iracema MP Calderon, MD, Phd, Study Director — Department of Gynecology and Obstetrics of Botucatu Medical School - São Paulo State University/UNESP. Botucatu, Brazil
Locations (1):
- Department of Gynecology and Obstetrics of Botucatu Medical School - São Paulo State University/UNESP, Botucatu, São Paulo, Brazil